CLINICAL TRIAL: NCT04685486
Title: Virtual Reality for Pain Management in Burn Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1610017629
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: Virtual Reality; Pain Management; Anxiety; Depression
MeSH Terms: conditions — Pain; Agnosia; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Virtual reality-enhanced distraction using a portable head mounted display during panful events (such as wound dressing changes or physical therapy sessions) in addition to standard of care.
  Interventions: Other: Virtual Reality
- Treatment as Usual (No Intervention): Standard of care during painful event (such as wound dressing changes or physical therapy sessions).

INTERVENTIONS:
Other: Virtual Reality — Immersive and interactive game played through a portable head-mounted display as a distraction mechanism
  Arms: Virtual Reality

SUMMARY:
This study is a randomized proof-of-concept study to assess the efficacy of Virtual Reality (VR) vs standard of care in 50 adult patients in the New York Presbyterian Burn Unit. The participants who are randomized to receive the virtual reality intervention will also receive opioids, which is the standard of care and is known to be effective. Participants will be randomly assigned to two groups. The first group will receive VR during their painful procedure (e.g., wound dressing changes, physical therapy etc.) in addition to the standard of care. The other group will receive standard of care (and no VR).

ELIGIBILITY:
Inclusion Criteria:

* 8 years and older
* Patients with a burn injury and is in the Burn Unit at New York Presbyterian
* Awake, alert, ambulatory
* The burn comprises less than 15% total body surface area (TBSA)
* The patient does not require conscious sedation such as ketamine for staple removal or wound dressing changes
* The patient is able to give informed consent

Exclusion Criteria:

* Diagnosis of a cognitive disorder, psychotic disorder or bipolar I as determined by self-report from previous diagnosis
* Current opioid abuse

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | Peri-procedural: 30 minutes before to two hours after the painful event.
  Initial determination of the clinical efficacy of VR in reducing the total pain (determined by the subjective standard 0-10 pain scale) where 0 = no pain and 10 = worst pain.
Change in narcotic dose | Peri-procedural: 30 minutes before to two hours after the painful event.
  Dose of narcotics needed peri-procedure

SECONDARY OUTCOMES:
Change in narcotic dose | Day 1 of hospitalization to last day of hospitalization (approximately 15 days)
  Determine if the one-time VR-distraction intervention reduces dose of analgesics for the day after the painful events and the remained of the post-procedure hospitalization
Change in anxiolytics dose | Day 1 of hospitalization to last day of hospitalization (approximately 15 days)
  Determine if the one-time VR-distraction intervention reduces anxiolytic dose after painful event
Change in Anxiety Symptoms | Peri-procedural: 30 minutes before to two hours after the painful event.
  Determined by visual analog scales (0-100) where 0 = no anxiety and 100 = worst possible anxiety.
Change in Depressive Symptoms | Peri-procedural: 30 minutes before to two hours after the painful event.
  Determined by visual analog scales (0-100) where 0 = no depression and 100 = worst possible depression.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No